CLINICAL TRIAL: NCT05974098
Title: Exploring the Impact of Illness Perceptions, Coping Strategies on Quality of Life in Paroxysmal Atrial Fibrillation Patients
Brief Title: Quality of Life Influencing Factors
Status: Completed | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Qu Shan, Head of the Department of Medical Psychology, Peking University People's Hospital
Other Study IDs: atrial fibrillation2023
Record Dates: First submitted 2023-07-20; First posted 2023-08-03 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Observation

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational study — This study intends to use correlation analysis and mediation analyses to assess the mediating effects of self-efficacy, coping, depression and anxiety on the quality of life of patients with paroxysmal atrial fibrillation.

SUMMARY:
Background: quality of life is impaired in patients with paroxysmal atrial fibrillation. The purpose of this study is to explore the mediating effects of self-efficacy, coping, depression, and anxiety on the quality of life of patients with paroxysmal atrial fibrillation. Methods: It is a cross-sectional study trial. This study aims to enroll 100 patients with paroxysmal atrial fibrillation. Illness perceptions (Brief Illness Perceptions Questionnaire; BIPQ), coping styles (Carver Brief-COPE scale; B-COPE), depression Patient Health Questionnaire-9 ,PHQ-9),anxiety (The Generalized Anxiety Disorder Questionnaire, GAD 7) and quality of life (12-item Short Form Health Survey,SF12) will be analysed. This study intends to use correlation analysis and mediation analyses to assess the mediating effects of self-efficacy, coping, depression and anxiety on the quality of life of patients with paroxysmal atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-75 years;
2. AF diagnosis, based on a 12-lead ECG and cardiologist-led examination following the 2016 ESC Guidelines for the Management of Atrial Fibrillation
3. paroxysmal AF diagnosis given by a cardiologist according to the conversion back to the normal sinus rhythm occurs spontaneously within a week
4. ability to read and write in Chinese.

Exclusion Criteria:

1. severe complications such as unstable coronary artery disease, heart failure with severe systolic dysfunction(ejection fraction≤35%)
2. AF soon after thoracic surgery;
3. malignant disease with a 1-year survival rate or a terminal illness diagnosis;
4. a diagnosed psychiatric condition that interfered with participation (including severe depression, bipolar disorder, psychotic illness of any type, dementia, acute suicidality, severe personality disorder)
5. participation in another study
6. cognitive impairment interfering with their ability to participate in the study

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients are from the Department of Cardiology and Department of Psychiatry, a comprehensive tertiary hospital in China. All patients who are interviewed provided written informed consents.
Sampling Method: Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
The 12-item Short Form Health Survey (SF-12) | Quality of life was measured at the start of the study，Up to 24 weeks
  The 12-item Short Form Health Survey (SF-12) is a 12-item, multipurpose short-form survey that is used to measure generic HRQoL (derived from the SF-36). The findings are weighted and summed to produce clearly interpretable scales for a participant's physical and mental well-being26. SF-12 is divided into two domains: the physical component summary (PCS) and the mental component summary (MCS). Each domain scores from 0 to 100, with higher scores indicating a better health status. The SF-12's PCS and MCS scores are based on the norms of a broad population in the United States of America, with a mean of 50

CONTACTS AND LOCATIONS:
Locations (1):
- Shan Qu, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Minjie Z, Zhijuan X, Xinxin S, Shan Q. Mediating effect of coping strategy and psychological status between illness perception and quality of life among patients with atrial fibrillation: a cross-sectional study. BMC Cardiovasc Disord. 2024 Sep 19;24(1):504. doi: 10.1186/s12872-024-04176-4. PMID 39300328